CLINICAL TRIAL: NCT04915781
Title: Tobacco Use and Incidence of SARS-CoV-2 Infection in the Finnish General Population
Brief Title: Tobacco Use and COVID-19 Incidence in the Finnish General Population
Acronym: Tobrisk-CoV
Status: Completed | Type: Observational
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Karolinska Institutet (Other); Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: THL/713/6.00.00/2021
Record Dates: First submitted 2021-06-03; First posted 2021-06-07 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: SARS-CoV-2 Infection; Covid19
Keywords: Tobacco use; SARS-CoV-2; COVID-19; Epidemiology; Cohort Studies; Incidence
MeSH Terms: conditions — COVID-19; Tobacco Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tobacco users: Never smokers (reference group) will be compared with former smokers, occasional smokers and daily smokers. For FinSote 2018 and 2020, we will also compare never users of (1) smokeless tobacco (snus), (2) electronic cigarettes with and without nicotine or (3) nicotine replacement therapy products with respective former, occasional and daily users.
  Interventions: Other: Not applicable, this is an observational study

INTERVENTIONS:
Other: Not applicable, this is an observational study — Not applicable, this is an observational study

SUMMARY:
This is an observational study of participants in three general population health surveys (FinSote 2018, 2019, 2020) who are followed up until the incidence of SARS-CoV-2 infection or end of follow-up. The primary objective is to examine the association between tobacco use and the risk of SARS-CoV-2 infection in a general population sample in Finland.

DETAILED DESCRIPTION:
Tobacco use, as a leading risk factor of death and disability due to respiratory diseases, was expected to increase the risk of SARS-CoV-2 infection and COVID-19 deaths. Earlier epidemiological studies, however, showed that smokers were underrepresented among patients hospitalized due to COVID-19. The most recent meta-analysis has confirmed these early findings, showing that current smokers had lower risk of SARS-CoV-2 infection than never smokers (Relative risk 0.71, 95% Credible interval 0.61; 0.82). A majority of these studies are based on samples of hospitalized patients, tested population or specific population groups, which might not represent the general population. In addition, data on tobacco use has been primarily collected from electronic health records or retrospectively and therefore prone to misclassification and information bias.

A message of a protective effect of tobacco use could undermine public health efforts to curb its use and reduce the perception of harm in the general population. Studies with general population samples and prospective data collection are thus urgently needed.

The aim of the study is to examine the association between tobacco use and the risk of SARS-CoV-2 infection. We will explore several forms of tobacco use (smoking, moist smokeless tobacco and e-cigarettes) and investigate whether introducing a potential collider bias by adjusting for mediating risk factors (alcohol use, physical activity and obesity) could have explained earlier results. We will use data from a prospective cohort study of nationally representative health surveys in Finland linked to SARS-CoV-2 incidence data, which is less subject to collider and recall bias than previous case-control studies.

ELIGIBILITY:
Inclusion Criteria:

* Permanent residents of Finland
* Registered in the Population Register at the moment of sampling
* Aged 20 and over
* Participated in the FinSote surveys in 2018, 2019 or 2020

Exclusion Criteria:

* Temporary residents in Finland or tourists
* Age less than 20 years old
* Did not participate in FinSote surveys in 2018, 2019 and 2020

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Permanent residents in Finland aged 20 and over who participated in the FinSote surveys in 2018, 2019 and 2020. These are general population samples representative of the Finnish population. The sampling frame was the Population Register (in 2020 the Digital and Population Data Services Agency, created after the merge between the Population Register of Statistics Finland and local register offices), which includes all individuals residing permanently in Finland, including conscripts and people living in institutions.
Sampling Method: Probability Sample
Enrollment: 60872 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of SARS-CoV-2 infection | Baseline until SARS-CoV-2 infection or April 30, 2021
  Incidence is the detection of a new SARS-CoV-2 infection with RT-PCR or a COVID-19 syndrome diagnosed by a physician from baseline to April 30, 2021

CONTACTS AND LOCATIONS:
Overall Officials: Sakari Karvonen, PhD, Principal Investigator — Finnish Institute for Health and Welfare
Locations (1):
- Finland, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
Researchers can access individual data by contacting the Responsible Researcher at the Finnish Institute for Health and Welfare, Suvi Parikka, suvi.parikka [at] thl.fi.
  Information about FinSote surveys, including questionnaires, can be found in https://thl.fi/fi/tutkimus-ja-kehittaminen/tutkimukset-ja-hankkeet/finsote-tutkimus

REFERENCES:
- [Background] Simons D, Shahab L, Brown J, Perski O. The association of smoking status with SARS-CoV-2 infection, hospitalization and mortality from COVID-19: a living rapid evidence review with Bayesian meta-analyses (version 7). Addiction. 2021 Jun;116(6):1319-1368. doi: 10.1111/add.15276. Epub 2020 Nov 17. PMID 33007104
- [Background] Bar-Zeev Y. Commentary on Simons et al. Public health implications of the suggested association between nicotine, smoking and infection with SARS-CoV-2. Addiction. 2021 Jun;116(6):1369-1370. doi: 10.1111/add.15356. Epub 2020 Dec 25. No abstract available. PMID 33368844
- [Background] Griffith GJ, Morris TT, Tudball MJ, Herbert A, Mancano G, Pike L, Sharp GC, Sterne J, Palmer TM, Davey Smith G, Tilling K, Zuccolo L, Davies NM, Hemani G. Collider bias undermines our understanding of COVID-19 disease risk and severity. Nat Commun. 2020 Nov 12;11(1):5749. doi: 10.1038/s41467-020-19478-2. PMID 33184277
- [Background] Haddad C, Bou Malhab S, Sacre H, Salameh P. Smoking and COVID-19: A Scoping Review. Tob Use Insights. 2021 Feb 15;14:1179173X21994612. doi: 10.1177/1179173X21994612. eCollection 2021. PMID 33642886
- [Background] Tattan-Birch H, Marsden J, West R, Gage SH. Assessing and addressing collider bias in addiction research: the curious case of smoking and COVID-19. Addiction. 2021 May;116(5):982-984. doi: 10.1111/add.15348. Epub 2021 Jan 20. No abstract available. PMID 33226690
- [Background] van Westen-Lagerweij NA, Meijer E, Meeuwsen EG, Chavannes NH, Willemsen MC, Croes EA. Are smokers protected against SARS-CoV-2 infection (COVID-19)? The origins of the myth. NPJ Prim Care Respir Med. 2021 Feb 26;31(1):10. doi: 10.1038/s41533-021-00223-1. PMID 33637750
- [Background] Vardavas CI, Nikitara K. COVID-19 and smoking: A systematic review of the evidence. Tob Induc Dis. 2020 Mar 20;18:20. doi: 10.18332/tid/119324. eCollection 2020. PMID 32206052
- [Background] Jimenez-Ruiz CA, Lopez-Padilla D, Alonso-Arroyo A, Aleixandre-Benavent R, Solano-Reina S, de Granda-Orive JI. [COVID-19 and Smoking: A Systematic Review and Meta-Analysis of the Evidence]. Arch Bronconeumol. 2021 Jan;57:21-34. doi: 10.1016/j.arbres.2020.06.024. Epub 2020 Jul 25. Spanish. PMID 34629638
- See also: Description of the Tobrisk-CoV project — https://www.nordforsk.org/projects/addressing-smoking-paradox-etiology-covid-19-through-population-based-studies-tobrisk-cov

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT04915781/Prot_SAP_000.pdf